CLINICAL TRIAL: NCT01549925
Title: A Prospective Randomized Surgical Trial Comparing the Efficacy of LIGASURE Assisted Recto-Sigmoid Resection and Omentectomy Compared to Standard Surgical Resection in Women With Stage IIIC or Stage IVA Epithelial Ovarian Cancer
Brief Title: Surgical Trial Comparing LIGASURE Assisted Recto-Sigmoid Resection and Omentectomy Compared to Stand
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCI41380
Record Dates: First submitted 2012-03-06; First posted 2012-03-09 (Estimated); Results first posted 2016-01-28 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2015-12

CONDITIONS: Epithelial Ovarian Cancer
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- standard surgical resection (Other): standard surgical resection using clamps and surgical ligatures
  Interventions: Other: Standard Surgical resection
- LIGASURE (Active Comparator): Resection using the FDA-approved LIGASURE device during omentectomy and resection of the recto-sigmoid portion of the colon
  Interventions: Device: LIGASURE

INTERVENTIONS:
Other: Standard Surgical resection — standard surgical resection using clamps and surgical ligatures
  Arms: standard surgical resection
Device: LIGASURE — resection using the FDA-approved LIGASURE device during omentectomy and resection of the recto-sigmoid portion of the colon
  Arms: LIGASURE

SUMMARY:
The objective of this prospective randomized surgical trial is to evaluate whether the use of the LIGASURE surgical device during omentectomy and/or recto-sigmoid resection for women with ovarian cancer will reduce the surgical time compared to standard surgical resection using clamps and surgical ligatures.

DETAILED DESCRIPTION:
This research study is a prospective, randomized trial. Women who are suspected to have an early or late stage ovarian cancer during their preoperative evaluation will be potential study participants. Only patients with documented ovarian cancer by histologic examination at the time of the cytoreductive or staging surgery, and that are also undergoing omentectomy and/or recto-sigmoid colon resection will be eligible for participation. Patients who are eligible for participation and who are willing to participate will be randomized during the surgical procedure to standard surgical resection using clamps and surgical ligatures versus resection using the FDA-approved LIGASURE device during omentectomy and resection of the recto-sigmoid portion of the colon. The resection of these tissues will be performed as part of the usual surgical protocol for women with ovarian cancer and will not be done so unless the tissues are the sites of metastatic disease or if their removal would be performed for staging purposes.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be 18 years or older
* All patients who are suspected to have an early or late stage ovarian cancer during their preoperative evaluation will be potential study participants.
* Potential candidates must have signed an IRB-approved Informed Consent (University of Utah Informed consent if their surgery will be performed at the Huntsman Cancer Hospital, or Intermountain Health Care consent if the surgery is to be performed at LDSH or IMC.
* Only patients with documented ovarian cancer by histologic examination at the time of the cytoreductive or staging surgery, and that are also undergoing omentectomy and/or recto-sigmoid colon resection will be eligible for participation.

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-01; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Intermountain Health Care, Salt Lake City, Utah
  - Huntsman Cancer Institute, Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard Surgical Resection | LIGASURE
Started | 25 | 25
Completed | 25 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Surgical Resection | LIGASURE | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Customized [Number; unit: Participants]
  < 50 years | 1 | 7 | 8
  50-70 years | 16 | 13 | 29
  >70 years | 8 | 5 | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 25 | 50
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Surgical Time
Description: To evaluate whether the use of the LIGASURE surgical device during omentectomy and/or recto-sigmoid resection for women with ovarian cancer will reduce the surgical time compared to standard surgical resection using clamps and surgical ligatures
Time Frame: at time of surgery, up to 10 minutes
Measure: Mean (95% Confidence Interval); unit: SECONDS
Arm/Group | Standard Surgical Resection | LIGASURE
Number analyzed (Participants) | 25 | 25
SECONDS | 417 [378 to 455] | 338 [296 to 379]

ADVERSE EVENTS:
Arm/Group | Standard Surgical Resection | LIGASURE
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No